CLINICAL TRIAL: NCT02844517
Title: Clinical Acceptance of the Artificial Pancreas: the International Diabetes Closed Loop (iDCL) Trial Research Site Training Protocol
Brief Title: International Diabetes Closed Loop (iDCL) Trial: Research Site Training Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Jaeb Center for Health Research (Other); TypeZero Technologies, LLC (Industry); Tandem Diabetes Care, Inc. (Industry); DexCom, Inc. (Industry); Roche Diagnostic Ltd. (Industry)
Responsible Party: Principal Investigator, Stacey Anderson, Study Chair, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19068; UC4DK108483 (NIH)
Record Dates: First submitted 2016-07-21; First posted 2016-07-26 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Artificial Pancreas; Closed Loop Control; Continuous Glucose Monitor (CGM)
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Pancreas, Artificial

STUDY DESIGN:
Intervention Model Description: The objective of the study is for clinical staff to gain experience using the proposed artificial pancreas system named inControl and the inControl Cloud and assess 24/7 in-home usability prior to initiating a large randomized controlled trial. Study subjects will wear the study insulin pump and CGM for approximately 2-4 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Artificial Pancreas (Experimental): The primary outcome is a qualitative assessment of the system's suitability for use in a large-scale in-home clinical trial based on the results of the Technology Acceptance questionnaire and feedback from clinical staff.
  Interventions: Device: Artificial Pancreas

INTERVENTIONS:
Device: Artificial Pancreas — Subjects will be provided the Artificial Pancreas (AP) system which includes the inControl Diabetes Management Platform, a study insulin pump and continuous glucose monitor. This AP system is designed to help control blood sugar in people living with type 1 diabetes.
  Other Names: inControl Diabetes Medical Platform

SUMMARY:
The objective of the study is for clinical staff to gain experience using the proposed artificial pancreas system named inControl and the inControl Cloud and assess 24/7 in-home usability prior to initiating a large randomized controlled trial.

DETAILED DESCRIPTION:
Participation in this study will require 5 study visits over 2-4 weeks.

* Visit 1: screening/enrollment visit to assess study eligibility.
* Visit 2: continuous glucose monitor (CGM) training and initiation session based upon current or prior use of a CGM; if subject doesn't currently use a CGM, subject will be trained and may be asked to wear the CGM at home for 1 week.
* Visit 3: subjects will be taught how to use the study insulin pump.
* Visit 4: subjects will be trained on the use of inControl and wear it at home for 14 days.
* Visit 5: subjects will return study equipment and to complete questionnaire.

ELIGIBILITY:
Inclusion Criteria

1. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year and using insulin for at least 1 year
2. Use of an insulin pump for at least 6 months with established parameters for basal rate(s), carbohydrate ratio(s) and insulin sensitivity factor(s) for at least 3 months.
3. Age 14.0 to <75.0 years
4. HbA1c level <10.5% at screening
5. For females, not currently known to be pregnant. If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative serum or urine pregnancy test will be required for all premenopausal women who are not surgically sterile. Subjects who become pregnant will be discontinued from the study. Also, subjects who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
6. Have care partner committed to participating in all training activities, knowledgeable at all times of the participants location, and being present and available to provide assistance when the system is being used at night
7. Willingness, if using the closed-loop system, to stop closed-loop when taking acetaminophen and avoid closed-loop for at least 4 hours afterward
8. Willingness to suspend use of any personal CGM for the duration of the clinical trial once the study CGM is in use
9. Willingness to establish network connectivity on a daily basis either via local Wi-Fi network or via a study-provided cellular service
10. Investigator has confidence that the subject can successfully operate all study devices and is capable of adhering to the protocol
11. Currently using no insulins other than one of the following rapid-acting insulins at the time of enrollment: insulin lispro (Humalog), insulin aspart (Novolog), or insulin glulisine (Apidra)
12. Total daily insulin dose (TDD) less than 100 U/day

Exclusion Criteria

1. More than one episode of diabetic ketoacidosis (DKA) in the 6 months prior to enrollment
2. More than one episode of severe hypoglycemia involving seizure of loss of consciousness in the 6 months prior to enrollment
3. Medical need for chronic acetaminophen
4. Concurrent use of any non-insulin glucose-lowering agent (including GLP-1 agonists, Symlin, DPP-4 inhibitors, SGLT-2 inhibitors, biguanides, sulfonylureas and naturaceuticals).
5. Hemophilia or any other bleeding disorder
6. A condition, which in the opinion of the investigator or designee, would put the participant or study at risk
7. Participation in another pharmaceutical or device trial at the time of enrollment or during the study
8. Employed by, or having immediate family members employed by TypeZero Technologies, LLC

Ages: 14 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome is a qualitative assessment of the system's suitability for use in a large-scale in-home clinical trial based on the results of the Technology Acceptance questionnaire and feedback from clinical staff. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boris P. Kovatchev, PhD, Principal Investigator — University of Virginia Center for Diabetes Technology; Stacey M. Anderson, MD, Study Chair — University of Virginia Center for Diabetes Technology
Locations (10):
- United States (7):
  - William Sansum Diabetes Center, Santa Barbara, California
  - Stanford University, Stanford, California
  - Barbara Davis Center, University of Colorado, Aurora, Colorado
  - Harvard University (Joslin Diabetes Center), Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Mt. Sinai, New York, New York
  - University of Virginia Center for Diabetes Technology, Charlottesville, Virginia
- University of Montpellier, Montpellier, France
- University of Padova, Padua, Italy
- Academic Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Not yet determined